CLINICAL TRIAL: NCT07226622
Title: Prescreening Study to Identify Potential Participants for a Clinical Study in Wilson Disease (WD) Due to the ATP7B p.H1069Q or p.R778L Mutations
Brief Title: Prescreening Study to Identify Potential Wilson Disease Participants for Gene-Editing Clinical Trial
Status: Recruiting | Type: Observational
Sponsor: Prime Medicine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Prime-0211
Record Dates: First submitted 2025-10-22; First posted 2025-11-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-10

CONDITIONS: Wilson Disease
Keywords: Hepatolenticular Degeneration; Liver Diseases; Genetic Diseases, Inborn; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Metabolism, Inborn Errors; Metal Metabolism, Inborn Errors; Metabolic Diseases; Nutritional and Metabolic Diseases
MeSH Terms: conditions — Hepatolenticular Degeneration; Liver Diseases; Genetic Diseases, Inborn; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Metabolism, Inborn Errors; Metal Metabolism, Inborn Errors; Metabolic Diseases; Nutritional and Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with at least 1 allele with the ATP7B p.H1069Q or p.R778L mutation

SUMMARY:
The aim of this study is to inform and improve future clinical trials in Wilson Disease (WD) by better understanding how patients with WD are living with and managing the disease, and by identifying key factors that shape their decisions to participate in clinical research.

DETAILED DESCRIPTION:
This will be a multi-region, multi-site, prescreening study for individuals with WD. Eligible participants must have a clinical history consistent with WD. p.H1069Q or p.R778L mutation are eligible for this study. Participants who do not have a known genotype at enrollment may have their ATP7B gene sequenced while on study, with the approval of the study Medical Monitor. Participants who have previously received liver transplant or gene therapy for WD are excluded.

This study will enroll up to approximately 30 participants aged 18 and above, at least 15 of whom must have at least 1 ATP7B p.H1069Q allele. Participants must meet all inclusion criteria and none of the exclusion criteria to be eligible for the study. Each participant will have a blood sample collected to evaluate total serum ceruloplasmin and ceruloplasmin oxidase. For participants who have at least 1 ATP7B allele with the p.H1069Q or p.R778L mutation, chart review will be conducted to collect relevant medical history information, and the participant will be asked to complete a survey to evaluate their interest in and attitudes towards gene editing for WD. Study participants will receive no study mandated therapeutic interventions but will continue to receive standard of care (SOC) for the treatment of WD. The expected duration of participation for each participant is approximately 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Wilson Disease (WD) as determined by the following criteria:

  1. An established clinical diagnosis of WD
  2. Genetic analysis confirming the presence of biallelic pathogenic variants at ATP7B, at least one of which is EITHER p.H1069Q OR p.R778L OR Participants without a confirmed genetic diagnosis may enroll only with explicit approval from the Medical Monitor

Exclusion Criteria:

1. Prior history of gene therapy, liver transplantation, hepatocyte (cellular) transplantation, or active listing for liver transplantation
2. For individuals with known ATP7B genotype: individual does not have at least 1 ATP7B allele with either the p.H1069Q or p.R778L mutation.
3. Significant neurological conditions within the prior 12 months which may impact participant safety or participation in the study, including ability to complete study requirements or procedures as outlined in the clinical study protocol.
4. In patients with psychiatric involvement, current or fluctuant clinical instability with new or changing diagnoses or substantial medication regimen changes in the past 12 months that could limit their participation, in the opinion of the Investigator.
5. History of cirrhotic decompensation within the past year.
6. Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the participant or would preclude the participant from successful study completion, including participant unable or unwilling to comply with the protocol requirements.
7. Current participation in an investigational study for the treatment of WD.
8. Prior or active malignancy or myeloproliferative disorder (excluding Stage 1 or lower, fully treated/excised malignant and pre-malignant disease of the skin, cervix or colon. Additionally, any other malignant and pre-malignant disease that the Investigator in consultation with the treating oncologist and study Medical Monitor deem has been fully treated/excised for > 5 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of Wilson Disease, at least 15 of whom have the p.H1069Q allele.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Gene Editing Interest & Attitudes Survey | From enrollment to the end of study 90 days
  This is a survey created by Prime Medicine. Survey answers are reported on both a scale and in open-ended response; the purpose of the survey is to better understand the patient's disease experience, current treatment and adherence, copper in diet and lifestyle, and gauge interest in a gene editing clinical study. No calculations with score values will be conducted.

SECONDARY OUTCOMES:
Distribution of serum ceruloplasmin levels | From enrollment to end of study 90 days
  The serum ceruloplasmin concentration will be measured once in all participants at a central laboratory using an oxidase activity-based assay.
Mutational landscape among adults with a clinically confirmed diagnosis of WD | From enrollment to end of study 90 days
  Targeted sequencing of ATP7B will be performed in participants whose index diagnosis of WD did not require diagnostic genetic testing
WD-related health characteristics | From enrollment to the end of study 90 days
  Targeted review of the available medical record will be performed and key health characteristics will be recorded and assessed in aggregate. A list of WD-related past medical history will be compiled. This will include all liver, neurological and psychiatric medical history categorized using MedDRA.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - University of California Davis Health, Sacramento, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medicine, Ann Arbor, Michigan
  - American Research Corporation, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
No plans to make IPD available to other researchers